CLINICAL TRIAL: NCT03518736
Title: Does Timing Matter? Efficacy of Parent Provided, Therapist Supported, Motor and Cognitive Intervention for Infants Born Very Preterm in the First Months of Life
Brief Title: Does Timing Matter? Supporting Play, Exploration, and Early Developmental Intervention
Acronym: TimeSPEEDI2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Stacey Dusing, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM20013026; FP00007043 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Preterm Infant; Cerebral Palsy
MeSH Terms: conditions — Premature Birth; Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Infants randomly assigned to this arm will not receive any study intervention but will continue with any intervention in the community recommended by their health care team.
- SPEEDI_Early (Experimental): Infants randomly assigned to this arm will participate in the SPEEDI intervention starting in the hospital and lasting for 4 months. This intervention includes 10 visits with a physical therapist and parent working together to advance an intervention program and 12 weeks of parent daily intervention.
  In addition they will continue with any intervention in the community recommended by their health care team.
  Interventions: Behavioral: Supporting Play Exploration and Developmental Intervention (SPEEDI)
- SPEEDI_Late (Experimental): Infants randomly assigned to this arm will participate in the SPEEDI intervention starting at 4 months post baseline or approximately 3 months after discharge from the hospital. This intervention includes 10 visits with a physical therapist and parent working together to advance an intervention program and 12 weeks of parent daily intervention.
  In addition they will continue with any intervention in the community recommended by their health care team.
  Interventions: Behavioral: Supporting Play Exploration and Developmental Intervention (SPEEDI)

INTERVENTIONS:
Behavioral: Supporting Play Exploration and Developmental Intervention (SPEEDI) — Physical Therapy intervention
  Arms: SPEEDI_Early; SPEEDI_Late

SUMMARY:
Infants born very preterm (≤28 weeks of gestation) are at high risk of having developmental disabilities including cerebral palsy, coordination impairments, attention deficit and learning disabilities. Impairment including reduced postural control, movement variability, visual motor skills, and motor learning are common during the first months of life and are associated with later developmental disabilities. However, infant born very preterm rarely receive evidence based therapeutic intervention in the first months of life when basic science and animal intervention studies suggest the greatest efficacy. Barriers to enrollment in services delay the onset of services and delivery models rarely support targeted preventative intervention or enhanced parent engagement during in the transition from the neonatal intensive care unit (NICU) to home.

Targeted intervention supporting postural control and motor learning in the NICU have resulted in short term motor gains. Interventions that enhance parent's ability to read their infant's cues and provide engagement opportunities improve maternal mental health and infant social and cognitive outcomes in the short-term. The purpose of this randomized clinical trial is to evaluate the efficacy of an intervention that combines evidence based motor intervention and parent engagement to enhance the parent's ability to provide daily motor and cognitive opportunities resulting in improved motor and cognitive outcomes.

Supporting Play Exploration and Development Intervention (SPEEDI) uses guided participation to empower parents in reading infant's behavioral cues, identifying ideal times for interaction, and enriching the environment and learning opportunities. Parents participate in 5 session in 3 weeks while learning principles of engagement, readiness for interaction, and to provide early motor and cognitive learning opportunities. Parents provide 20 minutes of motor and cognitive play based enrichment daily for 12 weeks with bi-weekly physical therapist support. The parent is empowered to determine the infant's current abilities and advance the activities to the "Just Right Challenge" throughout the 12 weeks, likely continuing after the intervention.

The efficacy of SPEEDI will be assessed during delivery at 2 time point; the transition from the NICU to home (around the infant's due date) and at 3-4 months of adjusted age (after the infants due date). Ninety infants will be randomly assigned to a Usual Care group, SPEEDI_Early, or SPEEDI_Later group. Group differences will be assessed in developmental outcomes on the motor and cognitive scales of the Bayley Scales for Infant and Toddler Development as well as the Early Problem Solving Indicator and Gross Motor Function Measure at the end of each intervention period, 12 and 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* All infants born very preterm (˂29 weeks of gestation) and cared for in the Neonatal Intensive Care Unit at the Children's Hospital of Richmond (CHoR) at Virginia Commonwealth University (VCU) or University of Virginia Hospital (UVa) will be offered an enrollment if they meet the following inclusion criteria.

  1. Infants must be medically stable, off ventilator support by 42 weeks of gestation
  2. live within 60 miles of either hospital (which are 75 miles apart). Early Intervention services in Virginia.
* A parent or LRA will also be enrolled in the study. Inclusion criteria for the adult is that they speak English and will be a caregiver for the enrolled infant.

Exclusion Criteria:

* Exclusion criteria include diagnosis of a genetic syndrome or unstable medical condition beyond 42 weeks of gestation.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Bayley Scaled of Infant and Toddler Development Cognitive and Gross Motor Scaled Scores | 6 months
  Scales scores for the cognitive and gross motor scales each have a mean of 10 and a standard deviation of 3. Higher scores are better.

SECONDARY OUTCOMES:
Assessment of Problem Solving in Play | 6 months
  This play based assessment of early problem solving skills quantifies the frequency of 5 behaviors
Gross Motor Function Measure (GMFM) | 6 months
  This is a measure of motor abilities that is sensitive to change for children with motor impairments. The GMFM-item set version will be used along with the Gross Motor Ability Estimator software to calculate a score on the GMFM-66.
Test of Infant Motor Performance (TIMP) | 3 months
  This is measure of motor abilities and selective motor control in infants less than 4 months of adjusted age or past their due date. The raw will be used to show change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Dusing, PT, PhD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Dusing SC, Burnsed JC, Brown SE, Harper AD, Hendricks-Munoz KD, Stevenson RD, Thacker LR, Molinini RM. Efficacy of Supporting Play Exploration and Early Development Intervention in the First Months of Life for Infants Born Very Preterm: 3-Arm Randomized Clinical Trial Protocol. Phys Ther. 2020 Aug 12;100(8):1343-1352. doi: 10.1093/ptj/pzaa077. PMID 32329778